CLINICAL TRIAL: NCT01540877
Title: A Human Experimental Model for Neuropathic Pain Using Combined Application of Capsaicin and Local Anesthetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Christoph Maier, Prof. Dr. med., Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HypCap
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2012-02-29 (Estimated); Status verified 2012-02

CONDITIONS: Ipsi- and Contralateral Hypoesthesia
MeSH Terms: interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Capsaicin application (Experimental): application of 0.6%
  Interventions: Procedure: Application of capsaicin 0.6%
- Local anesthetics application (Experimental): application of EMLA
  Interventions: Procedure: Application of local anesthetics (EMLA plaster)
- Combined application of 1. capsaicin 2. local anesthetics (Experimental): application of 1. capsaicin 0.6% and 2. EMLA
  Interventions: Procedure: Application of 1 capsaicin 0.6% and 2. EMLA
- Combined application of 1. local anesthetics and 2. capsaicin (Experimental): application of 1. EMLA and 2. capsaicin 0.6%
  Interventions: Procedure: Application of 1. EMLA and 2. capsaicin 0.6%

INTERVENTIONS:
Procedure: Application of capsaicin 0.6% — topical application of 0.6% capsaicin on the volar forearm
  Arms: Capsaicin application
Procedure: Application of local anesthetics (EMLA plaster) — topical application of EMLA on the volar forearm
  Arms: Local anesthetics application
Procedure: Application of 1 capsaicin 0.6% and 2. EMLA — topical application of 1. 0.6% capsaicin and 2. EMLA on the volar forearm
  Arms: Combined application of 1. capsaicin 2. local anesthetics
Procedure: Application of 1. EMLA and 2. capsaicin 0.6% — topical application of 1. EMLA and 2. 0.6% capsaicin on the volar forearm
  Arms: Combined application of 1. local anesthetics and 2. capsaicin

SUMMARY:
Main of the present study was to develop a model of concomitant C-fibre block and sensitization eliciting spontaneous pain as well applying topical capsaicin and local anesthetics (LA) to examine the sensory alterations after combined C-fiber block and sensitization in both different application orders (sensitization of blocked C-fibers and block of sensitized C-fibers), compared to each of both mechanisms alone. Thereby, we expect stronger sensory changes during the combined substance application than during the monoapplication. We expect also contralateral sensory alterations mirroring the changes on the intervention site after the combined capsaicin and LA application, being stronger than after sensitization alone absent after C-fiber block alone.

ELIGIBILITY:
Inclusion Criteria:

* healthy subject, older than 18 years, provided written informed consent

Exclusion Criteria:

* insufficient comprehension of the German language, history of severe internal, neurological or dermatological diseases, substance abuse, manifest psychiatric diseases, chronic and acute pain, any medication intake (except contraceptives in females) regularly or on demand during the last 14 days before study inclusion and during the study period, hypersensitivity to lidocaine or other amide-type anesthetics, hereditary or acquired methemoglobinemia, pregnancy, nursing, abnormal sensory profile in the quantitative sensory testing (QST) with side-to-side differences beyond the normal range at baseline and participation in clinical trials during the last month.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-04; Primary Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
grade of the ipsi- and contralateral hypoesthesia | 6 months

SECONDARY OUTCOMES:
area of the ipsi- and contralateral hypoesthesia | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pain Medicine, Bochum, Germany

REFERENCES:
- [Derived] Enax-Krumova EK, Pohl S, Westermann A, Maier C. Ipsilateral and contralateral sensory changes in healthy subjects after experimentally induced concomitant sensitization and hypoesthesia. BMC Neurol. 2017 Mar 23;17(1):60. doi: 10.1186/s12883-017-0839-9. PMID 28335745